CLINICAL TRIAL: NCT04730375
Title: Evaluation of the Effect of Different Doses Dexmedetomidine Infusion on Lung Mechanics and Oxygenation in Obese Patients Undergoing Laparoscopic Cancer Surgeries: A Randomized Controlled Trial
Brief Title: Evaluation of the Effect of Different Doses Dexmedetomidine Infusion on Lung Mechanics and Oxygenation in Obese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Mohammed Abdelfattah Abdelwadod, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2007-50109
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Obesity; Drug
MeSH Terms: conditions — Obesity | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: The study include 2 equal groups, each group is 35 patients: Group A(N=35) dexmedetomidine is infused intraoperative after intubation at dose of (1μg/Kg LBW) bolus, followed by 0.5μg/Kg/hour continuous infusion till the end of surgery and Group B(N=35) dexmedetomidine is infused intraoperative after intubation at dose of (0.5μg/Kg LBW) bolus, followed by 0.3μg/Kg/hour continuous infusion till the end of surgery.
Who Masked: Participant, Care Provider
Masking Description: Randomization is done using computer generated sequence. Concealment will be achieved by opaque envelope
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ( Group A) (Active Comparator): : Group A(N=35) dexmedetomidine is infused intraoperative after intubation at dose of (1μg/Kg LBW) bolus, followed by 0.5μg/Kg/hour continuous infusion till the end of surgery
  Interventions: Drug: Dexmedetomidine Injection [Precedex]
- (Group B) (Active Comparator): Group B(N=35) dexmedetomidine is infused intraoperative after intubation at dose of (0.5μg/Kg LBW) bolus, followed by 0.3μg/Kg/hour continuous infusion till the end of surgery.
  Interventions: Drug: Dexmedetomidine Injection [Precedex]

INTERVENTIONS:
Drug: Dexmedetomidine Injection [Precedex] — two different doses dexmedetomidine bolus then maintenance infusion till end of surgeries and evaluation of lung mechanics and oxygenation

SUMMARY:
• The objective of this study is to evaluate the effect of different doses of dexmedetomidine infusion intraoperative on lung mechanics and oxygenation regarding PaO2/Fraction of inspired oxygen), Intraoperative oxygenation, lung compliance (static and dynamic), dead space, and PaCO2,heart rate, mean arterial blood pressure in obese patients undergoing laparoscopic cancer surgeries

DETAILED DESCRIPTION:
Dexmedetomidine is a selective agonist of α2receptorswhose tendency to α2 receptors is eight times more than that of clonidine. It also has powerful sedative, analgesic, anti-inﬂammatory, and organ protective properties. dexmedetomidine has favorable respiratory effects in humans. The effects of dexmedetomidine on oxygenation and lung mechanics had been investigated in obstructive lung disease. Dexmedetomidine decreased dead space and improved both lung compliance and oxygenation in chronic obstructive pulmonary disease (COPD) patients undergoing lung cancer surgery. Morbidly obese patients are characterized by the high prevalence of restrictive lung disease.The study include 2 equal groups, each group is 35 patients: Group A(N=35) dexmedetomidine is infused intraoperative after intubation at dose of (1μg/Kg LBW) bolus, followed by 0.5μg/Kg/hour continuous infusion till the end of surgery and Group B(N=35) dexmedetomidine is infused intraoperative after intubation at dose of (0.5μg/Kg LBW) bolus, followed by 0.3μg/Kg/hour continuous infusion till the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60years
* Obese patients BMI>25 Kg/meter square
* Patients undergoing laparoscopic cancer surgery.

Exclusion Criteria:

* Heart failure
* Arrhythmias
* Severe liver or kidney impairment
* Patients with forced expiratory volume in 1 sec (FEV1)/FVC < 70%
* Heart block

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2021-01-30 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Oxygenation by the end study drug infusion | baseline and end of surgery
  PaO2/Fraction of inspired oxygen

SECONDARY OUTCOMES:
lung compliance | baseline and end of surgery
  static
lung compliance | baseline and end of surgery
  dynamic

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed abdel wadod, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Nataional Cancer Instituite, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided